CLINICAL TRIAL: NCT06704334
Title: The Study of Ginkgo Leaf Dropping Pills and Huperzine a Injection Combined with Median Nerve Electrical Stimulation in the Treatment of Cognitive Impairment After Brain Injury
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wanbangde Pharmaceutical Group Co., LTD (Industry)
Collaborators: Ganzhou City People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-03-06
Record Dates: First submitted 2024-04-30; First posted 2024-11-26 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Impairment After Brain Injury
MeSH Terms: interventions — huperzine A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Median nerve electrical stimulation group (Experimental): The optimal median nerve electrical stimulation treatment was given
  Interventions: Other: Median nerve electrical stimulation treatment
- Huperzine A injection + median nerve electrical stimulation group (Experimental): Huperzine A injection can be administered before median nerve electrical stimulation to improve the therapeutic effect of electrical stimulation.
  Huperzine A injection: intramuscular injection, 1ml,0.2mg once a day, the course of treatment was 7 days.
  Interventions: Other: Median nerve electrical stimulation treatment; Drug: Huperzine A injection
- Huperzine A injection + median nerve electrical stimulation + Ginkgo leaf dropping pill group (Experimental): Huperzine A injection can be administered before median nerve electrical stimulation to improve the therapeutic effect of electrical stimulation. After the end of the electrical stimulation treatment, ginkgo biloba dropping pills were given as long-term administration to maintain the therapeutic effect.
  Huperzine A injection: intramuscular injection, 1ml,0.2mg once a day, the course of treatment was 7 days.
  Ginkgo leaf dropping pills: Oral, each pill weighs 63mg, 5 pills/time, 3 times/day, the course of treatment is 3 months.
  Interventions: Other: Median nerve electrical stimulation treatment; Drug: Huperzine A injection; Drug: Ginkgo leaf dropping pill

INTERVENTIONS:
Other: Median nerve electrical stimulation treatment — Median nerve electrical stimulation is an electrical stimulation therapy in which the electrode is placed at the median nerve point 2cm above the carpal wrinkles on the palmar surface of the wrist joint. Generally, the right median nerve is used for electrical stimulation. Electrical stimulation improves cognitive function by stimulating neurons in the brain and improving information transmission between neurons. When electrical current stimulates the brain, it can increase the activity level of neurons and promote the signal transmission between neurons. Its mechanism of action includes the regulation of neurotransmitter acetylcholine, thereby enhancing cognitive function.
Drug: Huperzine A injection — intramuscular
  Arms: Huperzine A injection + median nerve electrical stimulation + Ginkgo leaf dropping pill group; Huperzine A injection + median nerve electrical stimulation group
Drug: Ginkgo leaf dropping pill — oral
  Arms: Huperzine A injection + median nerve electrical stimulation + Ginkgo leaf dropping pill group

SUMMARY:
This study will conduct a single-center clinical trial to explore the initial therapeutic effect of ginkgo biloba dropping pills, huperzine A injection and median nerve electrical stimulation in patients with cognitive impairment.

DETAILED DESCRIPTION:
Specific experimental research methods were randomized, controlled, single-center, exploratory clinical study, through the treatment of ginkgo biloba dropping pills, huperzine A injection and median nerve electrical stimulation in patients with cognitive impairment, to observe the effects of their neuroprotection and cognitive function improvement.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old

  * Residual cognitive impairment due to brain injury

    * No previous history of brain-related diseases except this one

Exclusion Criteria:

* The patient had severe underlying disease and unstable vital signs

  * The patient was complicated with consciousness disorder and could not cooperate with cognitive function assessment ③ Allergic to drugs or contraindications in drug use ④ There are contraindications of median nerve electrical stimulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
to assess the MMSE score | baseline，Day10，Day90

SECONDARY OUTCOMES:
to assess the MoCA score | baseline，Day10，Day90
to assess the ADAS-cog score | baseline，Day10，Day90
to assess the HAMD score | baseline，Day10，Day90
to assess the HAMA score | baseline，Day10，Day90

CONTACTS AND LOCATIONS:
Locations (1):
- The Ganzhou City People's Hospital, Ganzhou, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No